CLINICAL TRIAL: NCT00290927
Title: Evaluation of Efficacy and Safety of HMR1964 Intensive Therapy in Subjects With Type 2 Diabetes Mellitus Not Optimally Controlled With Oral Hypoglycemic Agents (OHA); OHA Therapy Controlled, Open, Randomized, Parallel Group, Comparative (Superiority), 16-week, Multinational, Multicenter Study
Brief Title: Efficacy and Safety of Insulin Glulisine in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6168
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: HMR1964, insulin glulisine, Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — insulin glulisine

INTERVENTIONS:
Drug: insulin glulisine

SUMMARY:
* To evaluate the superiority in the efficacy of HMR1964 and OHA combination therapy as compared with OHA therapy.
* To evaluate the superiority in the efficacy of HMR1964 mono-therapy as compared with OHA therapy.
* To evaluate the safety of HMR1964.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with type 2 diabetes mellitus diagnosed at least one year prior to the study with a BMI < 30 kg/m2 , a HbA1C of > 8.0 - < 11.0% at screening
* Fasting serum C-peptide at screening > 0.7 ng/mL
* Subjects who have been on a stable regimen and at the following doses of SU for at least 8 weeks prior to signing informed consent
* Glibenclamide > 5 mg/day
* Glimepiride > 3 mg/day
* Gliclazide > 80 mg/day In addition to receiving the above mentioned SU agents, subjects may have been treated with a biguanide at a stable dose for at least 8 weeks prior to signing informed consent.
* Subjects willing to administer three HMR1964 injections per day immediately prior to meals for a 16 week

Exclusion Criteria:

* Subjects unwilling or incapable of receiving a starting dose of ≥ 0.2 IU/kg/day of HMR1964
* Subjects with the likelihood of requiring concomitant treatment during the study period with the following classes of drugs: additional OHA (including thiazolidinediones, α-glucosidase inhibitors, D-phenylalanine derivative) other than those specified in the study protocol, insulin preparations other than HMR1964, systemic corticosteroids, other investigational products
* Subjects with clinically relevant cardiovascular, hepatic, neurologic, endocrine diseases; and active cancer; or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* Subjects who are pregnant, breast feeding or wish to become pregnant during the study period
* Subjects with diabetic retinopathy who received surgical treatments (laser photocoagulation or vitrectomy) within 12 weeks prior to informed consent, who are expected to have these surgical treatments during the study period, or who were diagnosed newly proliferative diabetic retinopathy within 12 weeks prior to informed consent

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390
Dates: Start 2003-12

PRIMARY OUTCOMES:
Efficacy: change in HbA1C from baseline to endpoint (superiority of HMR1964 and OHA combination therapy as compared to OHA therapy, superiority of HMR1964 mono-therapy as compared to OHA therapy)
Safety of HMR1964

SECONDARY OUTCOMES:
change in HbA1C from baseline to week 16,consecutive change in HbA1C every 4 wks,plasma glucose parameters, symptomatic hypoglycemia (comparison of HMR1964 intensive therapy, mono-or OHA combination therapy, with OHA therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Masayoshi KOYAMA, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Tokyo, Japan

REFERENCES:
- [Result] Kawamori R, Iwamoto Y, Kadowaki T, Iwasaki M, Kim SW, Woo JT, Baik SH, Yoon KH. Effects of insulin glulisine as mono- or add-on therapy in patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2009 Sep;11(9):900-9. doi: 10.1111/j.1463-1326.2009.01088.x. Epub 2009 Jul 13. PMID 19614946